CLINICAL TRIAL: NCT06763692
Title: Early Feasibility Study of Low-Intensity Focused Ultrasound (LIFU) Neuromodulation in Patients with Parkinson's Disease
Brief Title: Low Intensity Focused Ultrasound for Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ali Rezai (Other)
Responsible Party: Sponsor-Investigator, Ali Rezai, Director RNI, West Virginia University
Organization: West Virginia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RNI_NMD_PD
Record Dates: First submitted 2025-01-03; First posted 2025-01-08 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- LIFU Neuromodulation (Experimental)
  Interventions: Device: LIFU Neuromodulation

INTERVENTIONS:
Device: LIFU Neuromodulation — Subjects will undergo a single LIFU of the target brain region

SUMMARY:
This study is a prospective, single-center, single-arm early feasibility study, to establish safety and tolerability of LIFU for neuromodulation in patients with parkinson's Disease

DETAILED DESCRIPTION:
The primary objective is to evaluate the safety, feasibility and tolerability of LIFU as an adjunct neuromodulatory treatment for Parkinson's Disease

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant females aged 45 - 80 years at time of enrollment.
* Able and willing to give informed consent.
* Diagnosis of probable idiopathic Parkinson's disease by United Kingdom Parkinson's Disease
* Clinical diagnosis based on the Level II Movement Disorder Criteria and an FAQ less than or equal to 9.
* If on medication for the treatment of PD, or other medications for any other underlying medical conditions, must be on a stable dose for ≥4 weeks prior to Screening.
* Willing to not receive DBS or any other approved or experimental surgical or medical therapy for PD during the study period.
* Males and non-pregnant females aged 45 - 80 years at time of enrollment.
* Able and willing to give informed consent.
* Diagnosis of probable idiopathic Parkinson's disease by United Kingdom Parkinson's Disease
* Clinical diagnosis based on the Level II Movement Disorder Criteria and an FAQ less than or equal to 9.
* If on medication for the treatment of PD, or other medications for any other underlying medical conditions, must be on a stable dose for ≥4 weeks prior to Screening.
* Willing to not receive DBS or any other approved or experimental surgical or medical therapy for PD during the study period.

Exclusion Criteria:

* Unable to undergo MR-imaging because of non-MR compatible implants (e.g., pacemakers, medication pumps, aneurysm clips, metallic prostheses (including metal pins and rods, heart valves or cochlear implants), shrapnel fragments, permanent make-up or small metal fragments in the eye that welders and other metal workers may have), or if candidates are uncomfortable in small spaces (have claustrophobia).
* Active or chronic infection/inflammation
* Acute or chronic hemorrhages, specifically any lobar microbleeds with GRE and no siderosis or macro hemorrhages
* Tumor/space occupying lesion anywhere in the brain
* Participants who are unable or unwilling to lay flat and tolerate the required prolonged stationary position during treatment (approximately 2-3 hours).
* Participants with more than 30% of the skull area traversed by the sonication pathway are covered by scars, scalp disorders (e.g., eczema), atrophy of the scalp, or implanted objects in the skull or the brain.
* Participants with known unstable cardiac status or uncontrolled hypertension
* History of any clinically significant neurological disorder or procedure (e.g., brain surgery for Parkinson's disease, tumors, uncontrolled epilepsy, or any others deemed clinically significant by the investigator).
* Participant who has had deep brain stimulation or a prior stereotactic ablation of the basal ganglia, or thalamus.
* Currently participating in another clinical investigation with an active treatment arm or participated in any experimental therapy (drug or biologic or device) within 3 months prior to Screening.
* Use of any medications that, in the opinion of the Investigator, may contribute to cognitive impairment, put the participant at higher risk for AEs, or impair the participant's ability to perform cognitive testing or complete study procedures.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Treatment Emergent Adverse Events | baseline and day 7, 30 and 90 after study procedure
  All adverse events that are related to LIFU will be assessed

SECONDARY OUTCOMES:
Effect of LIFU on visuospatial function, | baseline and day 7, 30 and 90 after study procedure
  prosaccade (PST) and antisaccade (AST) task